CLINICAL TRIAL: NCT04401059
Title: Synergistic Real-World Study and Evidence-based Medicine Evaluation of Elemene Combined With Tyrosine Kinase Inhibitors（TKIs）in the Treatment of Advanced Non-small Cell Lung Cancer (NSCLC): Prospective Study
Brief Title: Synergistic Effect of Elemene Plus TKIs Compared With TKIs in EGFR-mutated Advanced NSCLC：Prospective Study
Acronym: SELECT-2
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Tian Xie (Other)
Collaborators: LinkDoc Technology (Beijing) Co. Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Tian Xie, Professor, Hangzhou Normal University
Organization: Hangzhou Normal University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HangzhouNU-2
Record Dates: First submitted 2020-05-18; First posted 2020-05-26 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Carcinoma; Non-Small-Cell Lung Cancer; Adenocarcinoma
Keywords: Elemene; TKI; EGFR; Real-world study
MeSH Terms: conditions — Carcinoma; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma | interventions — elemene; aumolertinib; aflutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Elemene plus First or Third generation EGFR-TKIs (Experimental): Elemene Injectable Emulsion sequentially with Elemene Oral Emulsion plus First -generation EGFR-TKIs (Gefitinib,Erlotinib, Icotinib) or Third-generation EGFR-TKIs (including but not limited to Osimertinib, Almonertinib, Furmonertinib).
  Interventions: Drug: Elemene plus first or third generation EGFR-TKIs
- First or third generation EGFR-TKIs only (Active Comparator): First-generation EGFR-TKIs (Gefitinib,Erlotinib, Icotinib) or third-generation EGFR-TKIs (including but not limited to Osimertinib, Almonertinib, Furmonertinib).
  Interventions: Drug: First or third generation EGFR-TKIs

INTERVENTIONS:
Drug: Elemene plus first or third generation EGFR-TKIs — Elemene Injectable Emulsion: 20ml: 88mg, 6 injections each time, once a day, continuous intravenous drip for 5 days. Continue to use Elemene Oral Emulsion. For specific usage, refer to the drug label.
  Elemene Oral Emulsion: 20ml: 176mg, 1 dose each time, 3 times a day. Use the Elemene Oral Emulsions until the disease progresses, the intolerable toxicity, the patient withdraws from the study, or dies for any reason.
  First or third generation EGFR-TKIs: refer to the drug label.
  Other Names: H10960114, H20010338
  Arms: Elemene plus First or Third generation EGFR-TKIs
Drug: First or third generation EGFR-TKIs — refer to the drug label.
  Other Names: Gefitinib(Iressa,YiRuiKe), Erlotinib(Tarceva), Icotinib(Kaimeina), Osimertinib(Tagrisso), Almonertinib, Furmonertinib, etc.
  Arms: First or third generation EGFR-TKIs only

SUMMARY:
This is a nationwide, multicenter and prospective cohort study. The purpose of this study is to evaluate the synergistic effect and safety of Elemene plus TKIs in EGFR-mutated advanced non-small cell lung cancer.

DETAILED DESCRIPTION:
About 9.2%-45.8% of Chinese patients with Non-small cell lung cancer were positive for EGFR gene mutation. Gefitinib, Erlotinib, Icotinib, Afatinib showed efficacy superior to that of chemotherapy in the treatment of EGFR mutation positive advanced NSCLC, and lower rates of serious adverse events. However, after a median of 8 to 13 months of disease control, patients ultimately progress due to acquired resistance of EGFR-TKIs. Elemene, a chemotherapeutic isolated from the Chinese medicinal herb Rhizoma Zedoariae, has been shown to have a comprehensive anti-tumor effect and the potential effect on reversing drug resistance.

In this study, about 22 research centers will participate in. We planned to enroll 744 patients with advanced non-small cell lung adenocarcinoma who were positive for EGFR mutations. The dynamic random method will be adopted in this study. Patients will be randomly divided into the experimental group（Elemene plus first or third generation EGFR-TKIs), and control group (First or third generation EGFR-TKIs, only). The purpose of this study is evaluating the synergistic effect and safety of Elemene plus TKIs in EGFR-mutated advanced non-small cell lung cancer. We also try to analyze the correlation between molecular biomarkers and patient prognosis, including but not limited to drug-resistant genes and circulating tumor cells.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18.
2. Histologically or cytologically confirmed advanced non-small cell lung adenocarcinoma(stage IIIB~IV).
3. Patients with EGFR mutations (deletions in exon 19 and L858R in exon 21 of the EGFR gene), plan to receive First-generation EGFR-TKIs (Gefitinib, Erlotinib, Icotinib) or third generation EGFR-TKIs (including but not limited to Osimertinib, Almonertinib, Furmonertinib) monotherapy for the first time (patients who have been using first- or third-generation EGFR-TKIs for less than 28 days can be enrolled).
4. Patients positive for EGFR gene mutation (deletions in exon 19 and L858R in exon 21 of the EGFR gene), with disease progression after receiving chemotherapy can be enrolled.
5. Confirmed by investigators, tumor tissue can't be surgically excised.
6. No prior exposure to elemene injectable and/or oral emulsion within one month.
7. Prior exposure to other Chinese patent medicine with similar efficacy within one month. If more than one month, patients can be enrolled after a 30-day washout period (without continuing to use the above medications).
8. The participant must be capable of understanding and complying with the protocol and willing to sign a written informed consent document.

Exclusion Criteria:

1. Patients with any EGFR mutations other than 19DEL or 21L858R.
2. Accompanied by other active tumors. (Except for stable basal cell carcinoma after treatment， If metachronous tumors have been controlled, participating was allowed )
3. Exposure to First- or third-generation EGFR-TKIs combined treatment, for example, chemotherapy, anti-angiogenesis therapy.
4. Receiving radiotherapy or chemotherapy.
5. Pregnant or lactating women.
6. Allergic to Elemene.
7. Participating in other drug clinical trials.
8. Refuse to comply with the follow-up.
9. The researchers did not consider it appropriate to participate in this study for other reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 744 (Estimated)
Dates: Start 2020-11-09 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
PFS | Start of treatment until 1-year follow-up
  PFS was defined as the interval from the date of randomization to the date of the first evidence of disease progression or death, whichever occurs first. Disease progression was defined according to RECIST 1.1.

SECONDARY OUTCOMES:
ORR | Start of treatment until 1-year follow-up
  ORR was defined as the percentage of participants with the best overall response (BOR) of complete response (CR) or partial response (PR) based on RECIST 1.1.
DCR | Start of treatment until 1-year follow-up
  Disease Control Rate (DCR) = Complete Response (CR) + Partial Response (PR) + Stable Disease (SD) as defined by RECIST 1.1.
OS | Start of treatment until 1-year follow-up
  Overall survival (OS) was defined as the interval from the date of randomization to date of death from any cause, or the date of last known follow-up alive.
Incidence and severity of AE or SAE | Start of treatment until 30 days after the last treatment
  Any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.
  A serious adverse event (experience) or reaction is any untoward medical occurrence that at any dose: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, or is a congenital anomaly/birth defect
Incidence and severity of ADR or SADR | Start of treatment until 30 days after the last treatment
  All noxious and unintended responses to a medicinal product related to any dose should be considered adverse drug reactions.
  A SADR is a serious ADR according to the above criteria of SAE.

OTHER OUTCOMES:
Quality of life (QOL) | Start of treatment until 1-year follow-up
  Quality of Life (QOL) was measured using the European Organization for Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC QLQ-C30 + LC 13).
Karnofsky Performance Scale (KPS) | Start of treatment until 1-year follow-up
  KPS: Performance status were measured using Karnofsky Performance Scale (KPS)
Traditional Chinese Medical(TCM) symptoms score | Start of treatment until 1-year follow-up
  TCM symptom score: Traditional Chinese Medical symptoms were measured from these eight aspects: chest pain, oppression in the chest, blood stasis, shortness of breath, weakness, palpitations, dry mouth, vexation. Particular attention should be paid to chest pain and weakness.
Molecular biomarkers | Start of treatment until 1-year follow-up
  Including but not limited to drug-resistant genes and circulating tumor cells. Such as PD-L1、MSI-H/dMMR、TMB、HLA、POLE、POLD1、DDR、TP53、KRAS、BRCA2、PBRM1、MDM2/4、EGFR、ALK、PTEN、JAK1/2、DNMT3A、STK11.

CONTACTS AND LOCATIONS:
Overall Officials: Ziping Wang, PhD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (7):
- China (7):
  - Affiliated Hospital of Nantong University, Nantong, Jiangsu
  - Panjin Central Hospital, Panjin, Liaoning
  - Shuguang Hospital Affiliated to Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality
  - The Second People's Hospital of Yangcheng County, Jincheng, Shanxi
  - Sichuan Academy of Medical Sciences· Sichuan Province People's Hospital, Chengdu, Sichuan
  - Hangzhou Cancer Hospital, Hangzhou, Zhejiang
  - Peking University Cancer Hospital, Beijing

IPD SHARING:
Plan to Share IPD: Undecided